CLINICAL TRIAL: NCT02699619
Title: Undisplaced Femoral Neck Fractures Treated With 2 Hansson Pins Without Plate or 3 Hansson Pins Interlocked in a Plate (Pinloc) - A Randomized Controlled Trial Using Radiostereometry
Brief Title: Undisplaced Femoral Neck Fractures 2 Hansson Pins or 3 Pins Interlocked in Plate (Pinloc) Using RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Frede Frihagen, Consultant, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/191/REK SO B
Record Dates: First submitted 2016-01-20; First posted 2016-03-04 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Hip Fractures; Femoral Neck Fractures
Keywords: Undisplaced
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures | interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 Hansson pins without plate (Active Comparator): Patients with undisplaced femoral neck fractures operated with 2 isolated Hansson pins.
  Interventions: Device: 2 Hansson pins
- 3 Hansson pins interlocked in a plate (Active Comparator): Patients with undisplaced femoral neck fractures operated with 3 Hansson pins interlocked in plate (Pinloc).
  Interventions: Device: Pinloc

INTERVENTIONS:
Device: Pinloc — 3 hook pins interlocked in plate.
  Other Names: 3 hook pins interlocked in plate.
  Arms: 3 Hansson pins interlocked in a plate
Device: 2 Hansson pins — 2 isolated hook pins.(Without plate)
  Other Names: 2 isolated hook pins.
  Arms: 2 Hansson pins without plate

SUMMARY:
Femoral neck fractures represent about half of the hip fractures and are further divided into displaced and undisplaced fractures. Displaced femoral neck fractures are almost always treated surgically with arthroplasty. However there is an ongoing debate on which implant is superior for undisplaced fractures.

A novel implant design (Pinloc) has been developed by Swemac Innovation AB. While the original implant consisted of 2 isolated hook pins, the modified design consists of 3 titanium hook pins interlocked in an aluminum plate. Interlocking is a new principle of implant design and improves fixation and load transfer amongst the pins. The superiority of the modified design is so far only proven preclinically.

The role of the Pinloc in clinical use remains unclear. Investigators are planning a randomized controlled trial on undisplaced femoral neck fractures to establish a method for implanting the tantalum markers, to observe the fracture healing process and to further investigate the role of the Pinloc.

DETAILED DESCRIPTION:
Femoral neck fractures represent about half of the hip fractures and are further divided into displaced and undisplaced fractures. Displaced femoral neck fractures are almost always treated surgically with arthroplasty. However there is an ongoing debate on which implant is superior for undisplaced fractures.

A novel implant design (Pinloc) has been developed by Swemac Innovation AB. While the original implant consisted of 2 isolated hook pins, the modified design consists of 3 titanium hook pins interlocked in an aluminum plate. Interlocking is a new principle of implant design and improves fixation and load transfer amongst the pins. The superiority of the modified design is so far only proven preclinically. The role of the Pinloc in clinical use remains unclear.

A series of studies is now planned at Oslo University Hospital in collaboration with Diakonhjemmet Hospital in hope to further clarify this debate. The use of the Pinloc has been introduced in some regions (e.g. Norway, Sweden and Japan). The role of the Pinloc remains unclear and very little has been published on it's use, even though it is believed to be an important contributor of stability to the fixation.

Femoral neck fractures are mainly caused by a fall from own height in the elderly. The fractures are most often classified as displaced or not, using the simplified Garden classification. Several other classification systems also exist, but these have not been shown to be of reliable clinical usefulness. The ideal classification system should be easily applicable, reliable, and aid in treatment decision making and prognosis.

The treatment of femoral neck fractures comprise perioperative and operative modalities. The perioperative modalities consist among others of medical optimalization preoperatively, early rehabilitation and prevention of new fractures by treating osteoporosis and preventing new falls. The main scope of the current study will, however, be the operative modalities.

Surgery for undsiplaced femoral neck fractures is performed mainly with internal fixation on a traction table, using either screws, pins or a sliding hip screw (SHS), available in various designs from different manufacturers. The latest Cochrane review did not conclude on which implant is the superior.

Radiostereometry (RSA) is the most precise and accurate method to measure motion in vivo between different segments in orthopaedic research. To do so, radioopaque tantalum markers are implanted into the bone defining different segments. Stereoradiographs are performed over time to detect movement and monitor the healing (or non healing) process. This movement can be calculated both as translations and rotations. They are ideal to describe and compare the stability of fracture systems. RSA has been used successfully in earlier studies on fracture healing. Due to the high accuracy and precision, RSA yield reliable results with relatively small study-groups. Investigators plan to use RSA to measure fracture dislocation and time to healing in our studies. The study will be on the function of the Pinloc and it´s ability to prevent secondary dislocation in undisplaced femoral neck fractures. Investigators will utilize RSA for measurements during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* undisplaced femoral neck fractures
* able to walk independently, aids such as crutches or walker allowed
* able to consent
* fit for surgery with pins with or without plate

Exclusion Criteria:

* not willing or able to attain follow up
* previous fracture or surgery with retained metal work in the same hip
* concomitant disease that will shorten life expectancy (i.e. cancer, COPD)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in fracture displacement during healing measured with radiostereometry | Up to 52 weeks
  Will be measured by RSA postoperatively, before discharge and after 4, 8, 12, 24 and 52 weeks. Total displacement from first reading to the reading showing maximum displacement is the main outcome.

SECONDARY OUTCOMES:
Perioperative blood loss | 1 week
Time of surgery | 1 week
Eq5d | 52 weeks
  Health Related Quality of Life (Hrqol).
Eq5d | 26 weeks
  Hrqol.
Eq5d | 12 weeks
  Hrqol.
Eq5d | 4 weeks
  Hrqol.
Change in time to union as measured by RSA (cessation of motion) and radiographs | Will be examined at 4, 12, 26 and 52 weeks
  When RSA shows that no motion has happened between two time points the fracture will be regarded as healed at the former time point.
Change in time to union as measured by plain radiographs and clinical findings | Will be examined at 4,12, 26 and 52 weeks
  Composite endpoint: Healing defined by obliteration of fracture line radiographically and pain free weight bearing (except lateral pain from hardware), when this occurs the fracture will be considered healed.
Harris Hip Score | Up to 52 weeks
  Will be examined at 4,12, 26 and 52 weeks
Postoperative pain (NRS) while in hospital | 1 week
  Pain at mobilization (NRS) at discharge
Timed Up and Go test | 4 weeks
  Tug
Timed Up and Go test | 12 weeks
  Tug
Timed Up and Go test | 26 weeks
  Tug
Timed Up and Go test | 52 weeks
  Tug
Pain (NRS) | 4 weeks
  Maximum hip pain during the last week
Pain (NRS) | 12 weeks
  Maximum hip pain during the last week
Pain (NRS) | 26 weeks
  Maximum hip pain during the last week
Pain (NRS) | 52 weeks
  Maximum hip pain during the last week
Satisfaction with operated hip (NRS) | 4 weeks
  NRS
Satisfaction with operated hip (NRS) | 12 weeks
  NRS
Satisfaction with operated hip (NRS) | 26 weeks
  NRS
Satisfaction with operated hip (NRS) | 52 weeks
  NRS
Motion during healing as measured by radiostereometry. | Up to 52 weeks
  Will be measured by RSA postoperatively, before discharge and after 4, 12, 24 and 52 weeks.
Motion during healing as measured by plain radiographs. | Up to 52 weeks
  Will be measured by RSA postoperatively, before discharge and after 4,12, 24 and 52 weeks.
Reoperation for healing problems | 52 weeks
  Any additional surgery addressing healing problems or hardware failure
Mortality | 52 weeks
  Any reason

CONTACTS AND LOCATIONS:
Overall Officials: Frede Frihagen, PhD, Principal Investigator — Oslo UH
Locations (1):
- Orthopedic Center, Ulleval University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
International peer review journal